CLINICAL TRIAL: NCT00177866
Title: The Safety of Celecoxib (Celebrex) in Patients With Crohn's Disease
Brief Title: Safety of Celecoxib in Patients With Crohn's Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: We were unable to get additional funding to complete study.
Sponsor: University of Pittsburgh (Other)
Collaborators: Shadyside Hospital Foundation (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0312013
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2016-07-15 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-06

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A Placebo or Celebrex (Active Comparator): either placebo PO BID for the first eight weeks or Celebrex 200 mg PO BID for the first eight weeks
  Interventions: Drug: Celebrex
- B Placebo or Celebrex (Placebo Comparator): either placebo PO BID for the last eight weeks or Celebrex 200 mg PO BID for the last eight weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Celebrex — Celebrex 200 mg PO BID for the first 8 weeks, followed by a 1 week "washout period" then placebo PO BID for the remaining 8 weeks - or - placebo PO BID for the first 8 weeks, followed by a 1 week "washout period" then Celebrex 200 mg PO BID for the remaining 8 weeks.
  Other Names: Celecoxib (brand name)
  Arms: A Placebo or Celebrex
Drug: placebo — placebo PO BID for either the first eight weeks or the last eight weeks of the study.
  Arms: B Placebo or Celebrex

SUMMARY:
The investigators will select 60 people who are 18-70 years of age with Crohn's disease and randomly assign them to receive an 8-week trial of celecoxib and an 8-week trial of a placebo. There will be a 1-week interval or "wash-out" between trials when the participant does not take any study medication. The investigators will monitor the participants for 18 weeks after they start the medication and observe their Crohn's disease activity, assessing for flare-ups or exacerbations in the disease and other possible side effects of celecoxib. Based on these observations, a determination will be made by the investigators as to the safety of celecoxib. If celecoxib is found to be safe, then it may provide physicians with a medication that they can prescribe for people who have Crohn's disease and experience chronic pain from arthritis and arthralgia.

DETAILED DESCRIPTION:
Please refer to brief summary (above).

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age or less than 70 years of age
2. Confirmed diagnosis of Crohn's disease
3. Inactive disease (CDAI scores at baseline <150) or active disease (CDAI scores at baseline <200).

Exclusion Criteria:

1. Pregnant, nursing mothers and women of childbearing potential who are not using reliable contraception (i.e.: oral contraceptive pill [OCP], intrauterine device [IUD], Norplant)
2. Enrolled in any other study involving non-steroidal anti-inflammatory drug (NSAID) medications
3. NSAID use at time of study
4. Baseline moderate to severe Crohn's disease activity (CDAI > 200)
5. Current treatment of less than 6 months with mercaptopurine (6 MP) or immuran.
6. Treatment with current Crohn's medication for a period of less than 3 months
7. Surgery for Crohn's disease (within 1 month)
8. Known sensitivity to celecoxib, NSAIDs, or sulfonamides
9. History of gastritis, gastrointestinal bleeding, or peptic ulcer disease
10. Advanced kidney disease
11. Severe hepatic impairment
12. Subjects currently taking angiotensin-converting enzyme (ACE) inhibitors, furosemide, fluconazole, lithium, corticosteroids, and warfarin

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George L Arnold, MD, Principal Investigator — University of Pittsburgh

RESULTS

PARTICIPANT FLOW:
Recruitment Details: No results or publication, data destroyed due to age of study. Enrollment number retrieved from old IRB database and not from study records and cannot be verified.
Pre-assignment Details: No results or publication, data destroyed due to age of study.
Groups:
- Celebrex Followed by Placebo: either placebo PO BID for the first eight weeks or Celebrex 200 mg PO BID for the first eight weeks
  Celebrex: Celebrex 200 mg PO BID for the first 8 weeks, followed by a 1 week "washout period" then placebo PO BID for the remaining 8 weeks -
- Placebo Followed by Celebrex: Placebo PO BID for the first 8 weeks, followed by a 1 week "washout period" then Celebrex 200 mg PO BID for the remaining 8 weeks.
Period: Overall Study
Arm/Group | Celebrex Followed by Placebo | Placebo Followed by Celebrex
Started | 0 (No results or publication, data destroyed due to age of study.) | 0 (No results or publication, data destroyed due to age of study.)
Completed | 0 (No results or publication, data destroyed due to age of study.) | 0 (No results or publication, data destroyed due to age of study.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No results or publication, data destroyed due to age of study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Celebrex Followed by Placebo | Placebo Followed by Celebrex | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Crohn's Disease Activity Index (CDAI) Scores in Response to Treatment
Description: Change in Crohn's Disease Activity Index (CDAI) scores in response to treatment
Time Frame: completion of all study participants
Population: No results or publication, data destroyed due to age of study.
Arm/Group | Celebrex Followed by Placebo | Placebo Followed by Celebrex
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Short Inflammatory Bowel Disease Questionnaire (SIBDQ) Scores in Response to Treatment
Description: No results or publication, data destroyed due to age of study.
Time Frame: completion of all study participants
Arm/Group | Celebrex Followed by Placebo | Placebo Followed by Celebrex
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: No results or publication, data destroyed due to age of study.
Arm/Group | Celebrex Followed by Placebo | Placebo Followed by Celebrex
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No